CLINICAL TRIAL: NCT06522997
Title: A Phase 2b Dose-finding, Randomized, Placebo-controlled, Double-blind Study to Evaluate Efficacy and Safety of BAY 3283142 on Top of Standard of Care in Reducing Albuminuria in Patients With Chronic Kidney Disease
Brief Title: A Study to Learn About How Well BAY3283142 Works and Its Safety in Participants With Chronic Kidney Disease
Acronym: ALPINE 1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22040; 2023-505755-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: 5+1 parallel-arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, participants will be randomly assigned to receive study intervention. Investigators, participants and study personnel will remain blinded to each participant's assigned study intervention throughout the course of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Placebo Comparator): Placebo OD and sham titration after 14 days and after 28 days
  Interventions: Drug: Placebo
- Arm 2 (Experimental): BAY3283142 (dose 1) OD and sham titration after 14 days and after 28 days
  Interventions: Drug: BAY3283142
- Arm 3 (Experimental): BAY3283142 (dose 2) OD and sham titration after 14 days and after 28 days
  Interventions: Drug: BAY3283142
- Arm 4 (Experimental): BAY3283142 (dose 2) OD and uptitration to dose 3 OD after 14 days and sham titration after 28 days
  Interventions: Drug: BAY3283142
- Arm 5 (Experimental): BAY3283142 (dose 2) OD and uptitration to dose 3 OD after 14 days and to dose 4 OD after 28 days
  Interventions: Drug: BAY3283142
- Arm 6 (Experimental): BAY3283142 (dose 3) OD and uptitration to dose 5 OD after 14 days and sham titration after 28 days
  Interventions: Drug: BAY3283142

INTERVENTIONS:
Drug: BAY3283142 — Tablet, intake orally once daily
  Arms: Arm 2; Arm 3; Arm 4; Arm 5; Arm 6
Drug: Placebo — Matching with BAY3283142
  Arms: Arm 1

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD), CKD is a condition in which the kidneys' ability to work properly gradually decreases over time. A common sign of decreasing kidney function is the body losing too much of a protein called albumin in the urine. This condition is known as albuminuria. This can lead to a faster decline in kidney function. People who have high blood pressure and diabetes are more likely to have CKD and are at a higher risk of complications related to it.

BAY3283142 is a new drug that is being developed to treat people with CKD. It works by activating a protein that helps relax blood vessels and is thought to have beneficial effects in CKD.

In this study, researchers want to learn about how well different doses of BAY3283142 work when taken with standard treatment for CKD in reducing albumin in the urine of participants with CKD. They will compare the results of the change in the urine albumin-creatinine ratio (UACR) after 16 weeks for BAY3283142 with a placebo. A placebo looks like the study drug but does not have any medicine in it.

During the study, participants will take either of the following drugs:

* BAY3283142: Participants will take BAY3283142 as tablets by mouth.
* Placebo: Participants will take it in the same way as BAY3283142. Participants will continue taking the available standard treatment for CKD and other conditions they may have (for example, heart conditions and diabetes).

At the start of this study, the researchers will check the medical history and current medications of the participants. They will also perform a complete health check-up of all the participants. Researchers will take urine and blood samples from the participants at different time points to measure UACR and eGFR.

Participants will be divided equally into different groups. Only 1 group will receive placebo and the other groups will receive BAY3283142. Participants will take their assigned treatment for 16 weeks.

No one will know who receives which drug or dose of BAY3283142 during the study.

Participants will be in this study for around 23 weeks. This includes the time for screening before the start of treatment and follow-up with participants after treatment.

People can join this study if they:

* are 18 years of age or older and have been diagnosed with CKD
* have poor kidney function according to the eGFR test
* have abnormally high levels of albumin in the urine according to the UACR test
* have been taking certain drugs at a stable dose for management of high blood pressure, diabetes, kidney disease, etc. for at least 4 weeks before the start of the study

People cannot join this study if they:

* have low blood pressure
* have had a stroke or a heart attack, or were hospitalized because of heart failure in the 3 months before the start of the study
* have a serious liver disease
* have a kidney disease for which they need to take drugs that control the immune system The detailed requirements will be discussed between the study doctors and people considering joining this study.

Participants may or may not get the expected benefits of treatment with BAY3283142, but they will receive thorough medical check-ups during this study. These can help to improve individual treatment in the future and to identify unknown medical risks.

Some participants may experience medical problems during this study including pain and discomfort when blood samples are taken. Researchers will closely monitor and manage any medical problems the participants may have. They will not include people who should not take BAY3283142 due to known safety concerns.

The findings from this study may contribute to developing a new treatment option for people with CKD who have excess albumin in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age
* eGFR (Chronic Kidney Disease Epidemiology Collaboration formula) ≥20 and ≤75 mL/min /1.73 m^2 at Screening Note: One re-assessment of eGFR based on central laboratory values is allowed during the Screening period"
* UACR ≥200 mg/g and <3500 mg/g as determined by the geometric mean (as calculated by the central laboratory) of 3 morning void urine specimens obtained at Screening
* Treatment with the highest tolerated labeled dose of either angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blockers (ARB), unless such treatment is either not tolerated or contraindicated. Treatment dose must be stable dose for at least 4 weeks before Screening with no planned change of the therapy during the study
* If the participant receives any of the following treatments it should be stable for 4 weeks prior to Screening: sodium-glucose co-transporter-2 (SGLT2) inhibitor, finerenone, diuretics, endothelin-receptor antagonists, or glucagon-like peptide (GLP) receptor agonist

Exclusion Criteria:

* Systolic blood pressure (SBP) <100 mmHg at Visit 2 (baseline)
* Patients with a tendency for clinically relevant orthostatic hypotension at Screening and Visit 2 (baseline) as judged by the investigator
* SBP ≥160 mmHg, unless treated with ≥3 blood pressure lowering medications, at Screening or at Visit 2 (baseline)
* History of secondary hypertension other than CKD
* Hepatic impairment corresponding to Child-Pugh B or C or other significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis as indicated by e.g. AST or ALT >3x ULN or total bilirubin >2x ULN) at Screening
* Polycystic kidney disease, lupus nephritis or ANCA-associated vasculitis and any other kidney disease requiring immunosuppressive therapy within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 16 in the logarithm of urine albumin-creatinine ratio (UACR) | From baseline to Week 16

SECONDARY OUTCOMES:
Change from baseline over time in estimated glomerular filtration rate (eGFR) | From baseline to Week 16
Change from baseline over time in the logarithm of UACR | From baseline to Week 16
Number of participants with treatment-emergent adverse events (TEAEs), serious TEAEs, and TEAEs leading to permanent discontinuation of study intervention | From the first dose of study intervention up to 7 days after last intake of study intervention, up to 17 Weeks per each participant

CONTACTS AND LOCATIONS:
Locations (154):
- United States (25):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Balboa Research SMO+ - Chula Vista - West, Chula Vista, California
  - Balboa Research SMO+ - La Mesa, La Mesa, California
  - California Kidney Specialists - San Dimas, San Dimas, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Nova Clinical Research - Blake Medical Center, Bradenton, Florida
  - Renstar Medical Research - Deerwood Clinic, Ocala, Florida
  - Elixia Central Florida, Orlando, Florida
  - Florida Institue for Clinical Research, Orlando, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Research by Design, LLC | Chicago, IL, Chicago, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - Hinsdale, Hinsdale, Illinois
  - Triad Internal Medicine - Asheboro, Asheboro, North Carolina
  - Eastern Nephrology Associates - New Bern, New Bern, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Renal Disease Research Institute | Landry, Dallas, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Utah Kidney Research Institute | Salt Lake City, UT, South Salt Lake, Utah
  - Peninsula Kidney Associates - Hampton, Hampton, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Salem VA Medical Center - Cardiology, Salem, Virginia
  - Mendez Center For Clinical Research | Woodbridge, VA, Woodbridge, Virginia
- Argentina (8):
  - Centro de Investigaciones Metabolicas | Ciudad de Autonoma de Buenos Aires, Argentina, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Centro de Investigaciones Medicas Temperley | Buenos Aires, Argentina, Temperley, Buenos Aires
  - CEDIC Centro de Investigación Clínica | Buenos Aires, Argentina, CABA, Ciudad Auton. de Buenos Aires
  - Centro de Especialidades Medicas (Cemedic) | Cardiology Department, Villa Luro, Ciudad Auton. de Buenos Aires
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" (CEMIC), Buenos Aires
  - Centro Privado San Vicente Diabetes, Córdoba
  - Centro de Rehabilitacion Cardiovascular | San Luis, Argentina, San Luis
  - Fundacion Centro de Salud e Investigaciones Medicas | Santa Rosa, Argentina, Santa Rosa
- Belgium (6):
  - Epicura / Nephrology, Baudour
  - UZ Gent / Nephrology, Ghent
  - Jan Yperman Ziekenhuis / Nephrology, Ieper
  - UZ Brussel Nephrology, Jette
  - UZ Leuven / Nephrology, Leuven
  - AZ Delta / Nephrology, Roeselare
- China (18):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Capital Medical University (CMU) - Beijing Anzhen Hospital (BAH), Beijing
  - Peking University People's Hospital, Beijing
  - Sichuan University - West China Hospital, Chengdu
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital (SAMSPH), Chengdu
  - The First People's Hospital - Foshan, Foshan
  - Southern Medical University - Nanfang Hospital (Southern Hospital), Guangzhou
  - Jiangsu Province Hospital of Traditional Chinese Medicine (TCM), Nanjing
  - Renji Hospital Shanghai JiaoTong University of Medicine, Shanghai
  - Huadong Hospital, Affiliated to Fudan University, Shanghai
  - Shanxi Bethune Hospital, Taiyuan
- Greece (8):
  - General Hospital of Athens LAIKO, Athens
  - University General Hospital of Heraklion - Department of Paediatrics, Heraklion
  - University of Thessaly - General University Hospital of Larissa (UHL), Larissa
  - University Hospital of Ioannina (UHI), Nisos Ioanninon
  - University General Hospital of Patras | Nephrology Clinic, Pátrai
  - Hippokration General Hospital of Thessaloniki - 3rd Department of Paediatrics, Nephrology Unit', Thessaloniki
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
  - Hellenic Republic Ministry of Health & Welfare - General Hospital of Thessaloniki (George Papanikolaou), Thessaloniki
- India (6):
  - Mavani Research Center, Ahmedabad, Gujarat
  - Life Care Clinic (LifeCare Clinic & Research Centre (LCRC)), Bangalore
  - Madras Diabetes Research Foundation, Chennai
  - The Institute of Post Graduate Medical Education & Research (IPGMER) (SSKM Hospital), Kolkata
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi
  - Max Super Speciality Hospital, Saket (West Block), (A unit of Max Healthcare Institute Limited), New Delhi
- Italy (5):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Nefrologia, Dialisi e Trapianto, Bologna, Emilia-Romagna
  - ASST Papa Giovanni XXIII | Ospedale di Bergamo - SC Malattie Endocrine-Diabetologia, Bergamo
  - Azienda Ospedaliera Universitaria Gaetano Martino Messina - Nefrologia e Dialisi, Messina
  - Azienda Ospedaliero Universitaria di Modena_Policlinico - Nefrologia, Dialisi e Trapianto di Rene, Modena
  - Istituti Clinici Scientifici Maugeri S.p.A._Pavia - Nefrologia, Pavia
- Japan (24):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Fukui Prefectural Hospital, Fukui-shi, Fukui
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Hirohata Naika Clinic, Kitakyushu, Fukuoka
  - Jiyugaoka Yamada Internal Medicine Clinic, Obihiro, Hokkaido
  - Naka Kinen Clinic, Naka, Ibaraki
  - Komatsu Municipal Hospital, Komatsu, Ishikawa-ken
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Katta General Hospital, Shiroishi, Miyagi
  - Rinku General Medical Center, Izumisano, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Ehime Prefectural Central Hospital, Matsuyama
  - Nara Prefecture General Medical Center, Nara
  - Osaka General Medical Center, Osaka
  - Japanese Red Cross Saitama Hospital, Saitama
- Portugal (10):
  - Unidade Local de Saude Almada-Seixal | Hospital Garcia de Orta - Research Department, Almada, Lisbon District
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Carnaxide, Lisbon District
  - Unidade Local de Saude do Estuario do Tejo | Hospital de Vila Franca de Xira - Departamento de Formacao e Investigacao, Vila Franca de Xira, Lisbon District
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Centro Hospitalar do Medio Tejo | Unidade de Torres Novas - Nephrology Department, Torres Novas, Santarém District
  - Centro Clinico Academico Braga | Braga, Portugal, Braga
  - CHUC- Hospitais da Universidade de Coimbra - Nephrology Department, Coimbra
  - Centro Hospitalar Universitario de Lisboa Central | Hospital Curry Cabral - Nephrology Department, Lisbon
  - Associacao Protectora dos Diabeticos de Portugal | Departamento de Ensaios Clinicos, Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
- Singapore (6):
  - National University Hospital Medical Centre, Singapore
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - SingHealth Polyclinics - Pasir Ris, Singapore
  - Changi General Hospital, Singapore
- Slovakia (9):
  - Nemocnica Akademika L. Derera - UNB, Nefrologicka ambulancia, Bratislava
  - DIABEDA s.r.o., Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
  - B. Braun Avitum Nefrologicka Ambulancia | Galanta, Slovakia, Galanta
  - NephroCare | FMC-dialyzacne sluzby s.r.o. - Kosice, Košice
  - Univerzitna nemocnica Martin, Martin
  - Biodial | Puchov, Slovakia, Púchov
  - DIAB s.r.o, Rožňava
  - B. Braun Avitum Nefrologicka ambulancia | Sala, Slovakia, Šaľa
- Spain (10):
  - Gerencia de Gestion Integrada A Coruna | Department of Endocrinology and Nutrition, A Coruña, A Coruña
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Nephrology Department, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario de Valencia | Nephrology Department, Missing, Valencia
  - Hospital Quironsalud Barcelona | Internal Medicine Department, Barcelona
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Ferrol
  - Hospital Universitario Ramon Y Cajal - Medicina Interna, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz | Nephrology and Hypertension Department, Madrid
  - Hospital Universitario Nuestra Senora de Valme | Internal Medicine Department, Seville
  - Hospital Universitario Doctor Peset | Nephrology Department, Valencia
  - Hospital Universitario Y Politecnico La Fe - Nefrologia, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset - Njurkliniken, Gothenburg
  - Universitetssjukhuset i Linköping, Linköping
  - ProbareE Stockholm, Stockholm
  - Center For Diabetes, Academic Specialist Center, Stockholm
  - Akademiska sjukhuset (Uppsala University Hospital) - Njurkliniken, Uppsala
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Chi-Mei Medical Center, Liouyine, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (9):
  - Northern Care Alliance NHS Foundation Trust | Salford Royal Hospital - Nephrology, Salford, Manchester
  - University Hospitals Birmingham NHS Foundation Trust | Queen Elizabeth Hospital Birmingham - Clinical Research Facility, Birmingham
  - Cardiff and Vale University Health Board | University Hospital of Wales - Nephrology and Transplant, Cardiff
  - Epsom and St Helier University Hospitals NHS Trust | St Helier Hospital - Clinical Trials Unit, Carshalton
  - Hull University Teaching Hospitals NHS Trust | Hull Royal Infirmary - Academic Renal Research Department, Hull
  - Barts Health NHS Trust - Royal London Hospital - Nephrology, London
  - King's College Hospital NHS Foundation Trust | King's College Hospital - Renal Research Department, London
  - Manchester University NHS Foundation Trust | Manchester Royal Infirmary - Renal Care, Manchester
  - Lakeside Healthcare | Lakeside Surgery - Research Department, Northamptonshire

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers' patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22040